CLINICAL TRIAL: NCT06453083
Title: Prospective Randomized Trial Using Medrol Dose Packs for Post-Operative Pain Control
Brief Title: Medrol Dose Packs for Post-Operative Pain Control
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Joshua Klatt, Principle Investigator, University of Utah
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 155546
Record Dates: First submitted 2024-06-05; First posted 2024-06-11 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2025-01

CONDITIONS: Pain
Keywords: Adolescent Idiopathic Scoliosis (AIS); Steroid; Medrol; Placebo; Pain
MeSH Terms: conditions — Pain | interventions — Methylprednisolone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo tablets (Placebo Comparator): Encapsulated placebo tablets per day (dosage for day 1 following the surgery is 32mg, day 2 is 24mg, day 3 is 16mg, day 4 is 12mg, day 5 is 8mg and day 6 is 4mg.)
  Interventions: Drug: Placebo
- Medrol tablets (Experimental): Encapsulated steroid Medrol tablets (dosage for day 1 following the surgery is 32mg, day 2 is 24mg, day 3 is 16mg, day 4 is 12mg, day 5 is 8mg and day 6 is 4mg)
  Interventions: Drug: Medrol

INTERVENTIONS:
Drug: Placebo — Placebo tablets will be dispensed to the participants for 6-days.
  Arms: Placebo tablets
Drug: Medrol — Medrol tablets will be dispensed to the participants for 6-days.
  Other Names: methylprednisolone
  Arms: Medrol tablets

SUMMARY:
The investigators primary purpose of this study is to determine if the addition of a short course use of steroids following surgery for Adolescent Idiopathic Scoliosis (AIS) will improve post-operative pain management and shorten hospital length of stay.

DETAILED DESCRIPTION:
Post-operative pain control following AIS surgery is challenging. Sub-optimal pain management results in emotional distress and prolonged hospital length of stay. Previous studies have shown that a short course of steroids following spine surgery is safe and improves pain control. To better understand the effects of the addition of steroids to a routine pain management strategy, a randomized prospective study with and without steroids will determine the benefit, if any, to the addition of steroids to the investigators already used pain protocol.

ELIGIBILITY:
Inclusion Criteria:

* age range of 10-21
* received AIS surgery

Exclusion Criteria:

* participants out of the age range 10-21
* other forms of scoliosis (not AIS)

Ages: 10 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 57 (Actual)
Dates: Start 2023-01-13 (Actual); Primary Completion 2024-12-17 (Actual); Study Completion 2024-12-17 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) pain | Day 1, post Adolescent Idiopathic Scoliosis (AIS) surgery
  VAS pain score (0 no pain - 10 severe pain)
Visual Analog Scale (VAS) pain | Day 2, post (AIS) surgery
  VAS pain score (0 no pain - 10 severe pain)
Visual Analog Scale (VAS) pain | Day 3, post (AIS) surgery
  VAS pain score (0 no pain - 10 severe pain)
Visual Analog Scale (VAS) pain | Day 4, post (AIS) surgery
  VAS pain score (0 no pain - 10 severe pain)
Visual Analog Scale (VAS) pain | Day 5, post (AIS) surgery
  VAS pain score (0 no pain - 10 severe pain)
Visual Analog Scale (VAS) pain | Day 6, post (AIS) surgery
  VAS pain score (0 no pain - 10 severe pain)

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Klatt, M.D., Principal Investigator — University of Utah Orthopaedics
Locations (1):
- University of Utah Orthopaedic Center, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No